CLINICAL TRIAL: NCT03936790
Title: A Dose-response Study of Spinally Administered Ropivacaine Combined With a Fix Dose of Fentanyl for Elective Caesarean Section in Tall Parturients Under Combined Spinal-epidural Anaesthesia
Brief Title: Dose-response Study of Spinally Administered Ropivacaine for Caesarean Section in Tall Parturients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Paraskevi Matsota (Other)
Responsible Party: Sponsor-Investigator, Paraskevi Matsota, Associate Professor of Anesthesiology, 2nd Department of Anaesthesiology, School of Medicine, University of Athens, "Attikon" Hospital, Athens, Greece., Attikon Hospital
Organization: Attikon Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EBD866
Record Dates: First submitted 2019-04-26; First posted 2019-05-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Regional Anaesthesia; Cesarean Section
Keywords: cesarean section; combined spinal epidural anaesthesia; tall parturients; ropivacaine ED50 and MLAD
MeSH Terms: interventions — Ropivacaine; Fentanyl

STUDY DESIGN:
Intervention Model Description: The sequential distribution methodology (up-down sequential allocation)
Masking Description: Two anaesthetists are required to conduct the study: a study supervisor who sets the dose of the local anaesthetic for the next participant according to the sequential distribution algorithm and performs the technique and an anaesthetist responsible for recording the study parameters and for the clinical management of the parturient, blinded to the administered dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ropi_dosing (Other): The dose of ropivacaine for each parturient is determined by the response of the previous participant to a higher or lower dose according to the sequential distribution algorithm (up-down sequential allocation).
  Interventions: Other: Ropivacaine; Other: Fentanyl

INTERVENTIONS:
Other: Ropivacaine — In case of successful spinal anaesthesia, the dose of spinally administered ropivacaine will decrease by 0.375 mg for the next participant.In case of unsuccessful spinal anaesthesia, the dose of spinally administered ropivacaine will increase by 0.375 mg for the next participant.
Other: Fentanyl — A fix dose of fentanyl (15 mcg) will be co-administered spinally to all participants.

SUMMARY:
The main goal is to determine the optimum dose of ropivacaine, a local anaesthetic, that provides regional anaesthesia with no or minimum adverse effects (i.e. hypotension) when given spinally in healthy full term tall parturients scheduled to undergo caesarean section under combined spinal / epidural anaesthesia (CSEA). The participants' height threshold is based on a local anthropometric research, which included over 2000 people. According to the above research the investigators calculated the female height distribution and decided to include in the study those distributed in the upper quartile (75th to 99th percentile). The female height distribution of the upper quartile ranges from 167 to 184 cm.

Secondary objectives are adverse effects related to the anaesthetic technique (hypotension, discomfort, nausea, vomiting and pruritus), the speed of installation and the duration of the regional block (both sensory and motor), blood gas analysis of the newborn umbilical blood as well as newborn Apgar score and lastly the mothers' degree of satisfaction.

This is a prospective non randomized double-blinded trial in which a specific algorithm for the local anaesthetic dose will be adopted (up-down sequential allocation). A written informed consent will be required by all participants.

The perioperative management of all participants will follow standard clinical protocols.

The dose of ropivacaine for each parturient is determined by the response of the previous participant to a higher or lower dose according to the sequential distribution algorithm (up-down sequential allocation). Specifically, the dose of ropivacaine for each parturient (except for the first) will fluctuate by 0.375 mg depending on the success (decrease by 0.375 mg) or failure (increase by 0.375 mg) of the spinal anaesthesia of the previous parturient enrolled in the study. The local anaesthetic dose of the first participant will be determined by a short pilot study.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the dose-response relationship of subarachnoid (spinal) administered ropivacaine to healthy tall parturients scheduled to undergo elective caesarean section under combined subarachnoid / epidural anaesthesia (CSEA) with co-administration of a fixed dose of fentanyl. The dose-response relationship will be described by determining ED50 (Effective Dose 50) and MLAD (Minimum Local Anaesthetic Dose).

The height threshold of the participants is based on the study "National Anthropometric Research: Effectiveness of Ergonomic Measurements and Applications." By G. Scroumbelos, University of Piraeus. Based on the female height distribution of the previously mentioned Anthropometric Research, we chose the upper quartile (75th to 99th percentile) as an inclusion criterion in our study, which ranges from 167 to 184 cm.

Secondary objectives are spinal induced hypotension, speed of installation and duration of sensory and motor blockade, blood gas analysis of the umbilical circulation of the newborn, Apgar score of the newborn, adverse effects related to the anaesthetic technique (discomfort, nausea, vomiting, pruritus) and the degree of maternal satisfaction.

This is a prospective non randomized double-blinded trial in which a specific algorithm for the local anaesthetic dose will be adopted (up-down sequential allocation, described below). A written informed consent will be required by all participants.

The perioperative management of the participants follows standard clinical protocols. Specifically, conventional non-invasive monitoring consisting of five lead electrocardiography, pulse oximetry and automatic oscillometric cuff blood pressure is used. A low-dose spinal via the needle-through-needle combined spinal-epidural (CSE) technique is employed. With the patient in the sedentary position, the O3-O4 intervertebral space is located, followed by skin antisepsis and topical lidocaine infiltration. The loss of resistance technique is used in order to locate the epidural space.

The dose of ropivacaine for each parturient is determined by the response of the previous participant to a higher or lower dose according to the sequential distribution algorithm (up-down sequential allocation). Specifically, the dose of ropivacaine for each parturient (except for the first) will fluctuate by 0.375 mg depending on the success (decrease by 0.375 mg) or failure (increase by 0.376 mg) of the subarachnoid anaesthesia of the previous parturient enrolled in the study. A fix dose of fentanyl (15 mcg) will also be co-administered to all participants. The dose for the first participant will be tailored to the results of a preliminary empirical study of a small number of parturients not enrolled in the trial.

Success of subarachnoid anaesthesia. Successful subarachnoid anaesthesia is defined as (1) an adequate sensory block at the level of T6 or higher within 15 minutes of the spinal injection of the local anaesthetic and opioid, (2) no need for a supplementary dose (rescue dose) of local anaesthetic given epidurally for at least 50 minutes after subarachnoid infusion (maternal pain intensity measured by a Visual Analog Scale, VAS ≤ 3), (3) and the onset of surgery 15 minutes after spinal injection of the local anaesthetic and opioid. In the case of successful subarachnoid anaesthesia, the dose of the spinally administered ropivacaine for the next participant decreases by 0.375 mg.

Failure of subarachnoid anaesthesia. Unsuccessful subarachnoid anaesthesia is defined as (1) VAS > 3 and (2) the need for a rescue dose (ropivacaine 0.5% 3-5 ml given epidurally) once within 50 minutes after the spinal infusion. In this case, the dose of the spinally administered ropivacaine for the next participant increases by 0.375 mg.

Exclusion from the study. The participant will be excluded from the study if (1) VAS > 3 and (2) there is a need for two or more rescue doses administered epidurally within 50 minutes after subarachnoid infusion or (3) there is a need to switch to general anaesthesia. In this case, the same dose of ropivacaine is repeated for the next parturient enrolled in the study.

According to the study protocol, two anaesthetists are required to conduct the study: a study supervisor who sets the dose of the local anaesthetic for the next participant according to the sequential distribution algorithm (see above) and performs the technique and an anaesthetist responsible for recording the study parameters and for the clinical management of the parturient, blinded to the administered dose.

A specific algorithm will be employed for prevention and treatment of spinal induced hypotension, which includes co-hydration with crystalloids (10ml.kg-1) and use of vasopressors (phenylephrine and ephedrine). The algorithm is in agreement with the latest guidelines on the management of hypotension during caesarean section under spinal anaesthesia ("International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia." Anaesthesia. 2018).

Sample size and statistical analysis. The sequential distribution methodology described by Dixon and Massey (up-down sequential allocation) is applied for statistical analysis. Bibliographic data suggests that "up-down sequential allocation" gives reliable results with a sample size of 20 to 40 individuals.

Data analysis will be performed using the Stata ™ software (Version 10.1 MP, Stata Corporation, College Station, TX 77845, USA).

ELIGIBILITY:
Inclusion Criteria:

* ASA status I - II (ASA; American Society of Anesthesiologists)
* height: 167 to 184 cm
* age: 20 to 40 years old
* normal single pregnancy
* full term pregnancy (> 37 weeks)
* elective caesarean section.

Exclusion Criteria:

* refusal of the parturient, inability to communicate
* obesity (BMI> 35 Kg/m2)
* baseline maternal heart rate less than 60 or above 130 bpm
* high risk pregnancy (gestational hypertension, preeclampsia / eclampsia, gestational diabetes, multiple pregnancies)
* known or suspected foetal pathology (intrauterine growth retardation, poly- or oligohydramnios)
* history of clinically significant cardiovascular, pulmonary, hepatic, renal, neurological, psychiatric or metabolic disease
* active labour
* history of allergy in amidic anaesthetics or any of the drugs used in the trial
* contraindications for regional technique such as coagulation disorders, inflammation of the lumbar region, systemic sepsis
* dural puncture.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-02 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
ED50 of spinal ropivacaine administered to healthy tall parturients for cesarean delivery. | Two to three hours
  Median Effective Dose (ED50) of spinally administered ropivacaine (mg).
MLAD of spinal ropivacaine administered to healthy tall parturients for cesarean delivery. | Two to three hours
  Minimum Local Analgesic Dose (MLAD) of spinally administered ropivacaine (mg).

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi Matsota, MD, PhD, Principal Investigator — Associate Professor of Anaesthesiology, Second University Clinic of Anaesthesiology, Faculty of Medicine, University of Athens
Locations (1):
- 2nd Department of Anesthesiology, Attikon University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared starting 6 months after publication.

REFERENCES:
- [Background] Khaw KS, Ngan Kee WD, Wong EL, Liu JY, Chung R. Spinal ropivacaine for cesarean section: a dose-finding study. Anesthesiology. 2001 Dec;95(6):1346-50. doi: 10.1097/00000542-200112000-00011. PMID 11748390
- [Background] Siddiqui KM, Ali MA, Ullah H. Comparison of spinal anesthesia dosage based on height and weight versus height alone in patients undergoing elective cesarean section. Korean J Anesthesiol. 2016 Apr;69(2):143-8. doi: 10.4097/kjae.2016.69.2.143. Epub 2016 Mar 30. PMID 27066205
- [Background] Harten JM, Boyne I, Hannah P, Varveris D, Brown A. Effects of a height and weight adjusted dose of local anaesthetic for spinal anaesthesia for elective Caesarean section. Anaesthesia. 2005 Apr;60(4):348-53. doi: 10.1111/j.1365-2044.2005.04113.x. PMID 15766337
- [Background] Pace NL, Stylianou MP. Advances in and limitations of up-and-down methodology: a precis of clinical use, study design, and dose estimation in anesthesia research. Anesthesiology. 2007 Jul;107(1):144-52. doi: 10.1097/01.anes.0000267514.42592.2a. PMID 17585226
- [Background] Stroumpoulis K, Stamatakis E, Koutroumanis P, Loukeri A, Valsamidis D. Pencil-point needle bevel direction influences ED50 of isobaric ropivacaine with fentanyl in spinal anesthesia for cesarean delivery: a prospective, double-blind sequential allocation study. Int J Obstet Anesth. 2015 Aug;24(3):225-9. doi: 10.1016/j.ijoa.2015.03.005. Epub 2015 Mar 16. PMID 25936784
- [Background] Parpaglioni R, Frigo MG, Lemma A, Sebastiani M, Barbati G, Celleno D. Minimum local anaesthetic dose (MLAD) of intrathecal levobupivacaine and ropivacaine for Caesarean section. Anaesthesia. 2006 Feb;61(2):110-5. doi: 10.1111/j.1365-2044.2005.04380.x. PMID 16430561
- [Background] Geng ZY, Wang DX, Wu XM. Minimum effective local anesthetic dose of intrathecal hyperbaric ropivacaine and bupivacaine for cesarean section. Chin Med J (Engl). 2011 Feb;124(4):509-13. PMID 21362272
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733